CLINICAL TRIAL: NCT05514691
Title: A Study to Evaluate the Clinical Performance, Usability and Readability of the iStatis COVID-19 Ag Rapid Test Performed With Anterior Nasal Swabs
Brief Title: Evaluation of Clinical Performance and Usability of iStatis COVID-19 Ag Rapid Test at POC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CLS-011
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Virus Infection; COVID-19; Coronavirus Disease-19; COVID-19 Pandemic; SARS-CoV-2 Infection
Keywords: diagnostic kit; diagnostic devices; lateral flow device test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Enrolled subjects with anterior nasal swab are tested on both iStatis COVID-19 and RT-PCR.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Anterior nasal swab sample tested on iStatis Covid-19 Antigen Testing diagnostic device (Active Comparator): An anterior nasal swab was collected using the swab provided with the iStatis test kit and will be used for the iStatis Covid-19 Antigen Testing at the site.
  Interventions: Diagnostic Test: iStatis COVID-19 Ag Rapid Test
- Anterior nasal swab sample tested with RT-PCR (Active Comparator): Another anterior nasal swab sample was collected to be tested with RT-PCR at the central research laboratory.
  Interventions: Diagnostic Test: "COVID-19 RT-PCR Test EUA Number: EUA200011, Company: Laboratory Corporation of America ("Labcorp")

INTERVENTIONS:
Diagnostic Test: iStatis COVID-19 Ag Rapid Test — SARS-Cov-2 tests are performed on all appropriate swab samples from each subject enrolled as a comparator test to iStatis Rapid Test
  Arms: Anterior nasal swab sample tested on iStatis Covid-19 Antigen Testing diagnostic device
Diagnostic Test: "COVID-19 RT-PCR Test EUA Number: EUA200011, Company: Laboratory Corporation of America ("Labcorp") — The Labcorp COVID-19 RT-PCR or EURORealTime SARS-Cov-2 tests are performed on all appropriate swab samples from each subject enrolled as a comparator test to iStatis Rapid Test
  Arms: Anterior nasal swab sample tested with RT-PCR

SUMMARY:
A rapid point of care test for the detection of virus particles will be compared to the FDA approved EUA RT-PCR detection standard. The iStatis COVID-19 Ag Rapid Test is intended for rapid point-of-care detection of the SARS-CoV-2 nucleocapsid protein antigen.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the Clinical Performance of iStatis COVID-19 Antigen Test by untrained operators at Point of Care settings that meet requirements for CLIA waived tests.

Secondary Objective: To evaluate the performance of iStatis COVID-19 Antigen test around Limit of Detection Samples will be collected in CLIA Waived settings from approximately 200 subjects who present with or are referred for concerns about SARS-CoV-2. The goal is to collect a minimum of N=30 confirmed Covid-19 positive subjects and N=30 confirmed Covid-19 negative subjects of comparable ages, genders, and races.

Individual participation only includes sample collection and 1 day visit for the purpose of study

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing to sign verbal informed consent form
* Age 18 or older
* Subject is suspected case of COVID-19 by clinical criteria: a patient with acute respiratory tract infection (sudden onset of at least one of the following: cough, fever, shortness of breath, fatigue, decreased appetite, myalgia)
* Subjects with above mentioned symptom onset within the 7 days
* Participant is willing to provide two swabs - one anterior nasal swab sample for iStatis Test and another nasopharyngeal or nasal swab sample for comparator RT-PCR testing

Exclusion Criteria:

* Individuals who presented with 8 or greater days of COVID- 19 Related Symptoms, (Fever, Cough, Fatigue, Decreased Appetite, Shortness of Breath, Myalgia) or postdefervescence and/or convalescence
* Any reason as identified by the Principal Investigator at the participating site that could disqualify the subject from participation. The reason for exclusion was documented
* Subject withdraw consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Summary of the iStatis COVID-19 Ag test performance data compared to the comparator EUA RT-PCR test when all data from 4 POC/CLIA sites are combined. | 2 - 3 weeks
  The primary efficacy analyses will be analysis of relative positive percent agreement (PPA) and negative percent agreement (NPA) of the iStatis COVID-19 Antigen test results compared with the participant's RT-PCR results. The overall lower 95% confidence interval will be determined when:
  Positive Percent Agreement (PPA) = [TP / (TP + FN)] x 100, where
  * TP (true positive) is a positive iStatis test in agreement with prior positive RT-PCR test, and
  * FN (false negative) is negative iStatis test discordant with prior positive RT-PCR test.
  Negative Percent Agreement (NPA) = [TN / (TN + FP)] x100, where
  * TN (true negative) is a negative iStatis test in agreement with negative RT-PCR test, and
  * FP (false positive) is a positive iStatis test discordant with a negative RT-PCR test.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Centennial Medical Group, Elkridge, Maryland

IPD SHARING:
Plan to Share IPD: No